CLINICAL TRIAL: NCT06445231
Title: Implementation and Effectiveness of Screening Echocardiography Performed in Nursing Home: ECHOGER
Brief Title: Echocardiography in Nursing Home
Acronym: ECHOGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Directorate of Health Care Supply (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC22_0449
Record Dates: First submitted 2024-05-14; First posted 2024-06-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Heart Diseases; Heart Failure; Heart Valve Diseases
Keywords: Echocardiography; Nursing Home; Implementation; Heart Failure
MeSH Terms: conditions — Heart Diseases; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Nursing home randomization in 1:1 ratio between echocardiography and no-echocardiography
Masking Description: Not relevant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echocardiographic screening arm (Experimental): Participants from nursing homes allocated to echocardiographic screening group will benefit of one echocardiography at inclusion.
  Interventions: Diagnostic Test: Implementation of echocardiography in nursing homes
- Usual care (No Intervention): Participants from nursing homes allocated to no-screening group. Participants will be followed for medical management and care as usual.

INTERVENTIONS:
Diagnostic Test: Implementation of echocardiography in nursing homes — An ultrasound will be carried out in the EHPAD, the result of which will be interpreted by a cardiologist then sent to the establishment and the attending physician with instructions to follow.
  Arms: Echocardiographic screening arm

SUMMARY:
The study seeks to explore the implementation characteristics (acceptability, appropriateness, feasibility, adoption, fidelity, penetration, implementation cost and sustainability) of systematic echocardiography in nursing homes and its impact on rates of heart failure flare-up and unscheduled hospitalization at 12 months among included nursing homes.

DETAILED DESCRIPTION:
Open-label cluster randomized type 1 hybrid trial, with 2 parallel arms: nursing homes will be randomized in the interventional (echocardiography by sonographer) or non-interventional arms (usual care). In the interventional arm echocardiography will be proposed to all residents of the nursing home at baseline. Clinical management will be adapted to the result of echocardiography by the general practitioner, in accordance with the cardiologist. The main objective is to assess the impact at 12 months of the initial performance of a systematic simplified echocardiography on the rate of nursing home residents presenting with heart failure episode or cardiovascular pathology. The Primary endpoint is the number of nursing home residents presenting a heart failure episode or an unscheduled hospitalization for heart failure or other cardiovascular pathologies at 12 months.

Thirty nursing homes and 1050 residents will be included overall

ELIGIBILITY:
Inclusion Criteria :

Nursing homes residents with a life-expectancy estimated > 1 year, and able to participate to the study, giving an oral consent

Exclusion Criteria :

* no accessible to echocardiography
* closed unit (severe Alzheimer disease…)
* recent contagious disease such Covid (<15 days)
* no consent to participate
* no social security number

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Count of resident presenting a heart failure decompensation | 12 months
  Number of residents with heart failure flare (worsening of at least 1 NYHA class) or unplanned hospitalization for heart failure

SECONDARY OUTCOMES:
Presence of a clinically significative change in medical management and care in the month following ultrasound | 12 months
  A binary outcome will be constructed, based on the following algorithm: clinically significative change set to "yes" if a change in ongoing drug prescription is observed, and/or a cardiologist visit is planned, and/or a geriatrist visit is planned, and/or an hospitalization for clinical work-up is set, and/or a resume of the ultrasound is sent to the GP. Otherwise (all components set to "absent"), this outcome will be set to "None".

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LE TOURNEAU, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Yes